CLINICAL TRIAL: NCT02078258
Title: Attention Bias Modification Treatment for Major Depressive Disorder in Adolescents: A Randomized Controlled Trial
Brief Title: Attention Bias Modification Treatment for Major Depressive Disorder in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunan Normal University (Other)
Responsible Party: Principal Investigator, Wenhui Yang, Department of Psychology, Hunan Normal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2014-01-14; First posted 2014-03-05 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Major Depressive Disorder, Single Episode, Unspecified
Keywords: depression，adolescent，attention bias，modification
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Attentional bias modification training (Experimental): Attention bias modification training (ABMT) is a a variation of attention tasks to modify attentional biases, in which a probe always appears in the location of relatively positive stimuli after the two stimuli, one neutral and one emotional, were simultaneously presented.
  Participants complete 8 sessions (320 trials each with 20 minutes) over two weeks of neutral ABMT to shift attention toward neutral, in which a probe appeared in the location of neutral with 90% probability, and sadness-related with 10% probality. At a 9-week follow-up, participants completed 4 more sessions (480 trials each with 30 minutes)over two weeks of positive ABMT to shift attention toward positive words,in which a probe appeared in the location of 67% positive or 33% neutral.
  Interventions: Behavioral: ABMT
- Placebo control (Active Comparator): The placebo ABMT was identical to the active ABMT, but shifted toward neutral (50%) or sad (50%) stimuli equally often (i.e., 50/50 training).
  Interventions: Behavioral: ABMT

INTERVENTIONS:
Behavioral: ABMT — During a two-week period, 8 sessions of a modified dot probe task for attentional bias modification training (ABMT) condition, 8 sessions of a classic dot probe task for placebo training (PT) condition.

SUMMARY:
In this study, we test whether a two-week 8-session neutral attention bias modification (ABM) training and a two-week 4-session positive ABM could reduce depressive symptoms relative to placebo controls in adolescents with major depressive disorder at posttraining and follow-ups during one year.

DETAILED DESCRIPTION:
Depression is a common health problem in adolescents. Negative attentional bias has been theorized to play a critical role in the onset and maintenance of depression, suggesting that reduction of such biases may treat symptoms of depression. Recent studies have shown that attention bias modification(ABM) training could reduce depressive symptoms in both dysphoria and previously depressed adult patients.To test the effectiveness of ABM training on the treatment of depressive symptoms in depressed adolescents, we designed a randomized, double-blind, placebo controlled trial in adolescents with major depressive disorder(MDD).

ELIGIBILITY:
Inclusion Criteria:

* Meet the major depression disorder's criteria

Exclusion Criteria:

* bipolar disorder, schizophrenia or organic mental disorder;
* any concurrent psychotherapy;
* any concurrent psychotropic medication.

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2012-09; Primary Completion 2014-01 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Changes in depressive symptom number | baseline, 7-week, 6-month follow-up
  Depressive symptom accounts measured by Kiddie Schedule for Affective Disorders and Schizophrenia for School-Age Children.
Changes in depressive severity | baseline, 7-week, 6-month follow-up
  depressive severity measured by the construct interview of the Schedule for Affective Disorders and Schizophrenia for School-Age Children(K-SADS)

SECONDARY OUTCOMES:
Change of Self-report symptoms | baseline, 7-week, 6-, 12-month follow-up
  symptoms measured by the Center for Epidemiological Studies Depression Scale (CES-D), State-Trait Anxiety Inventory-Trait(STAI-T)，Rumination Response Style（RRS)，Suicidal Ideation Questionnaire（SIQ）
Diagnostic status of major depressive disorder | baseline, 7-week, 6-month follow-up
  Assessed by the diagnostic interview of the Schedule for Affective Disorders and Schizophrenia for School-Age Children

CONTACTS AND LOCATIONS:
Overall Officials: Wenhui Yang, Ph.D, MD., Study Director — Hunan Normal University
Locations (1):
- Department of Psychology, Hunan Normal University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
All data can be shared with other researchers
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: after the completion and forever
Access Criteria: Only for research

REFERENCES:
- [Result] Yang W, Zhang JX, Ding Z, Xiao L. Attention Bias Modification Treatment for Adolescents With Major Depression: A Randomized Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2016 Mar;55(3):208-18.e2. doi: 10.1016/j.jaac.2015.12.005. Epub 2015 Dec 23. PMID 26903254